CLINICAL TRIAL: NCT05092048
Title: Validation Value of the Questionnaire to Assess Health-related Quality of Life in Patients With CML
Brief Title: A Study for PRO of CML in Real Word
Acronym: Case-Only
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: xuna (Other)
Responsible Party: Sponsor-Investigator, xuna, professor, Nanfang Hospital, Southern Medical University
Organization: Nanfang Hospital, Southern Medical University (Other)
Other Study IDs: CML0922
Record Dates: First submitted 2021-09-22; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-09

CONDITIONS: CML (Chronic Myelogenous Leukemia)
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- CML patient: ≥18 years old CML patiente
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — PHQ-9 and GAD-7 questionnaire

SUMMARY:
Successful outcomes in CML require both prolonged adherence to oral TKI therapy by patients and careful monitoring of treatment responses by their physicians. Patient Reported Outcomes(PRO) assessment is important to facilitate decisions in the current treatment landscape of CML.

DETAILED DESCRIPTION:
1. Above 18 years of age.
2. Patient with confirmed diagnosis of Philadelphia chromosome positive and/or BCR-ABL positive chronic myeloid leukemia (CML).
3. Written informed consent.
4. Patients enrolled in investigational drug-trials or other type of clinical trials are also eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Above 18 years of age. Patient with confirmed diagnosis of Philadelphia chromosome positive and/or BCR-ABL positive chronic myeloid leukemia (CML).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Assess health-related Quality of Life and Symptom Burden in patients with chronic myeloid leukemia | 1 year
  Health-related quality of life (HRQOL) assessment in the current treatment landscape of chronic myeloid leukemia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, Nanfang Hospital, Southern Medical University,, Guanzhou, China

REFERENCES:
- [Derived] Chen H, Wen Y, Zeng Y, Lin L, Sun B, Zhu H, He H, Wang X, Zou W, Zheng C, Zheng L, Huang J, Pang L, Huang J, Zhang Y, Lin H, Liu Z, Zhu W, Wang Q, Zhou X, Liu X, Qu H, Liu Z, Du X, Xu N. Patient Versus Physician Perspective in the Management of Chronic Myeloid Leukemia During Treatment with Tyrosine Kinase Inhibitors. Oncol Ther. 2024 Mar;12(1):131-145. doi: 10.1007/s40487-023-00255-2. Epub 2023 Dec 16. PMID 38104036